CLINICAL TRIAL: NCT04314050
Title: Comparison of Different Strategies in Preventing Discomfort Due to Urine Catheter in Urinary Surgery
Brief Title: Comparison of Tramadol and Dexmedetomidine in the Prevention of Urinary Catheter Discomfort in Urinary Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Özkan Sipahioğlu, University of Health Sciences, Diskapi Yildirim Beyazit Training and Research Hospital, Department of Anesthesiology and Reanimation, Ankara Diskapi Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Urinery Catheter Discomfort
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Catheter Related Complication
Keywords: dexmedetomidine; tramadol; catheter-related bladder discomfort
MeSH Terms: interventions — Tramadol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tramadol (Active Comparator): 1,5 mg /kg tramadol will perform intraoperatively in 100 ml saline within 15 minutes at 30 minutes before surgery completed. In addition, 1 gr paracetamol will be given intraoperatively.
  Interventions: Drug: Tramadol
- dexmedetomidine (Active Comparator): 1 mcg/kg dexmedetomidine bolus will perform after anesthesia induction and followed by infusion of 0.5 mcg/kg/h until 30 minutes before surgery completed. In addition, 1 gr paracetamol will be given intraoperatively.
  Interventions: Drug: Dexmedetomidine
- control (Placebo Comparator): 1 gr paracetamol will perform intraoperatively
  Interventions: Other: control

INTERVENTIONS:
Drug: Tramadol — tramadol and paracetamol will perform
  Other Names: Contramal
  Arms: tramadol
Drug: Dexmedetomidine — dexmedetomidine and paracetamol will perform
  Other Names: precedex
  Arms: dexmedetomidine
Other: control — paracetamol will perform
  Arms: control

SUMMARY:
The investigators aimed to compare the effects of tramadol and dexmedetomidine, which are commonly used in anesthesia, on preventing catheter-related bladder discomfort.

DETAILED DESCRIPTION:
Urinary catheterization is an attempt frequently used in many surgeries, emergency services or intensive care units, especially urinary surgeries to facilitate urine output or evaluate urine output. However, as a result of urinary catheter application, most patients may develop some symptoms like pain, burning sensation and the urge to urinate constantly in the suprapubic region that the investigators call this catheter-related bladder discomfort (CRBD).

The incidence of CRBD can increase 47 to 90% in the postoperative period. The main reason of CRBD is involuntary contractions caused by muscarinic receptors, especially type 3 (M3) receptors. Therefore, antimuscarinic drugs are used to prevent and treat CRBD. Studies have shown that many drugs such as ketamine, tolterodine, oxybutynin, gabapentin, pregabalin, butylscopolamine, tramadol, dexmedetomidine are effective in preventing CRBD. Their common feature is antimuscarinic effects. However, no definitive conclusion could be reached for routine use, due to the low number of samples in the studies, surgical differences or some anticholinergic and sedative side effects. Additionally, oxybutynin, tolterodine, gabapentin, and pregabalin are only preoperatively administered orally. So more research is needed to find the ideal agent to prevent CRBD.

Tramadol is frequently used for moderate pain in surgeries. It is a centrally acting synthetic opioid analgesic that has an inhibitory effect on M1 and M3 muscarinic receptors. Tramadol has proven to be effective in reducing the severity and frequency of ICBR in intraoperative use. However, like other opioids, it can have side effects such as nausea-vomiting and sedation.

Dexmedetomidine is a selective alpha-2 adrenoceptor agonist that has analgesic, sympatholytic and sedative properties. In recent studies, it has been reported that dexmedetomidine is associated with the pathophysiology of CRBD by inhibiting type-3 (M3) muscarinic receptor which has beneficial effects in preventing CRBD in intraoperative use. Dexmedetomidine decreases the frequency of CRBD by 30%.

The first purpose of the study is to compare the effects of dexmedetomidine and tramadol on CRBD. Secondarily, the investigators aimed to compare them for their side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 70 years
* American Society of Anesthesiologists I or II
* Scheduled to undergo retrograde intrarenal surgery
* Scheduled to apply urinary catheter intraoperatively

Exclusion Criteria:

* History of bladder outlet obstruction (Bening prostatic hypertrophy)
* History of neurogenic bladder
* History of psychiatric illness
* Obese patient
* Patients whose urinary catheter cannot be inserted
* Patients who had previously urinary catheters

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — male patients
Enrollment: 135 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
the severity of CRBD | 0. hour
  none - mild- moderate- severe
the severity of CRBD | 1. hour
  none - mild- moderate- severe
the severity of CRBD | 3. hour
  none - mild- moderate- severe
the severity of CRBD | 6. hour
  none - mild- moderate- severe

SECONDARY OUTCOMES:
11-point numerical rating scale (NRS) | 24 hours
  11-point numerical rating scale for pain (0='no pain' and 10='worst pain possible pain') were explained

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Özkan Sipahioglu, specialist, Principal Investigator — Ankara Diskapi Research and Training Hospital
Locations (1):
- Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Hur M, Park SK, Yoon HK, Yoo S, Lee HC, Kim WH, Kim JT, Ku JH, Bahk JH. Comparative effectiveness of interventions for managing postoperative catheter-related bladder discomfort: a systematic review and network meta-analysis. J Anesth. 2019 Apr;33(2):197-208. doi: 10.1007/s00540-018-2597-2. Epub 2019 Jan 2. PMID 30603826
- [Background] Agarwal A, Yadav G, Gupta D, Singh PK, Singh U. Evaluation of intra-operative tramadol for prevention of catheter-related bladder discomfort: a prospective, randomized, double-blind study. Br J Anaesth. 2008 Oct;101(4):506-10. doi: 10.1093/bja/aen217. Epub 2008 Jul 24. PMID 18653496
- [Background] Kim HC, Lee YH, Jeon YT, Hwang JW, Lim YJ, Park JE, Park HP. The effect of intraoperative dexmedetomidine on postoperative catheter-related bladder discomfort in patients undergoing transurethral bladder tumour resection: A double-blind randomised study. Eur J Anaesthesiol. 2015 Sep;32(9):596-601. doi: 10.1097/EJA.0000000000000196. PMID 25485879
- [Background] Akca B, Aydogan-Eren E, Canbay O, Karagoz AH, Uzumcugil F, Ankay-Yilbas A, Celebi N. Comparison of efficacy of prophylactic ketamine and dexmedetomidine on postoperative bladder catheter-related discomfort. Saudi Med J. 2016 Jan;37(1):55-9. doi: 10.15537/smj.2016.1.14122. PMID 26739975
- [Result] Li S, Song L, Ma Y, Lin X. Tramadol for the treatment of catheter-related bladder discomfort: a randomized controlled trial. BMC Anesthesiol. 2018 Dec 20;18(1):194. doi: 10.1186/s12871-018-0659-5. PMID 30572837